CLINICAL TRIAL: NCT05838131
Title: A Clinical Trial to Explore the Safety and Efficacy of CT071 Injection in Patients With Relapsed/Refractory Multiple Myeloma or Primary Plasma Cell Leukemia
Brief Title: Study of CT071 Injection in RRMM or PPCL
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Juan Du, Chief physician, professor, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT071-CG7001
Record Dates: First submitted 2023-04-03; First posted 2023-05-01 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma; Primary Plasma Cell Leukemia
Keywords: multiple myeloma; primary plasma cell leukemia; CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells Infusion (Experimental): Biological: CART cells chimeric antigen receptor T cells
  Interventions: Drug: Experimental: CAR-T cells Infusion

INTERVENTIONS:
Drug: Experimental: CAR-T cells Infusion — Biological:
  chimeric antigen receptor T cells
  Other Names: Single Group Assignment

SUMMARY:
A Clinical Trial to Explore the Safety and Efficacy of CT071 injection in Patients with Relapsed/Refractory Multiple Myeloma or Primary Plasma Cell Leukemia

DETAILED DESCRIPTION:
This trial is a single-arm, open-label, dose-finding, first-in-human clinical trial. The main aim of this study is to preliminarily evaluate the safety and tolerability of CT071 after infusion, and explore the dose range of CT071 in patients with relapsed/refractory multiple myeloma or primary plasma cell leukemia, so as to determine the possible recommended therapeutic dose (RD).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the clinical trial; fully understand and are informed of this trial and sign the informed consent form; Willing to follow and able to complete all trial procedures;
2. Age ≥ 18 years, male or female;
3. Patients with multiple myeloma who have received at least three lines therapy for multiple myeloma (requires relapse, progression, non-response after treatment with at least 1 proteasome inhibitor and at least 1 immunomodulator.
4. Patients with primary plasma cell leukemia progressed after treatment with at least 1 regimen;
5. Progressive disease at the time of enrollment according to the IMWG consensus for myeloma or plasma cell leukemia;
6. Have any of the following evaluable conditions:

   1. Serum M-protein ≥ 5 g/L;
   2. 24-hour urine M-protein ≥ 200 mg;
   3. Abnormal serum free light chain (sFLC) ratio and affected FLC ≥ 100 mg/L in subjects with multiple myeloma who did not meet evaluable criteria for either serum or urine M-protein levels;
   4. Circulating plasma cells ≥ 5% (PCL subjects only);
7. Estimated survival > 12 weeks;
8. Eastern Cooperative Oncology Group (ECOG) score 0-2;
9. Subjects had adequate organ function.
10. Female subjects of childbearing potential must have a negative serum pregnancy test at screening, be willing to use a highly effective and reliable method of contraception within 1 year after receiving the trial treatment, and absolutely prohibit egg donation during the trial and within 1 year after receiving the trial treatment;
11. Male subjects, if sexually active with a female of childbearing potential, are willing to use a highly effective and reliable method of contraception for 1 year after receiving trial treatment. All male subjects are absolutely prohibited from donating sperm during the trial and for 1 year after receiving the trial treatment.

Exclusion Criteria:

1. Pregnant or lactating females;
2. Patients with a history of neurological disease, such as epilepsy, intracranial hemorrhage, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, memory impairment, spinal cord compression, psychiatric disease or any disease involving the central nervous system, or suspected central nervous system (CNS) metastasis;
3. Patients with other incurable malignant tumors within 5 years or at the same time, except for those with very low degree of malignancy;
4. Patients with active autoimmune diseases, including but not limited to psoriasis, rheumatoid arthritis, inflammatory bowel disease and other patients requiring long-term immunosuppressive therapy;
5. Received allogeneic stem cell transplantation within two years prior to screening;
6. Received autologous stem cell transplantation within 12 weeks prior to screening, or plan to receive autologous stem cell transplantation during the trial;
7. Any uncontrolled disease or disorder with important clinical significance investigator considered not applicable for the study;
8. Patients who had any uncontrolled active infection (defined as the presence of persistent signs or symptoms associated with infection that did not improve despite appropriate antiinfective treatment) or who required intravenous antiinfective agents (except for prophylactic treatment) within 4 weeks before apheresis. If there is clinical indications, investigators should consider screening EBV, CMV, and other related pathogenic microorganisms;
9. Major surgery within 2 weeks prior to screening, or planning to undergo major surgery within 4 weeks after trial treatment (excluding cataract and other surgery under local anesthesia);
10. Received treatment for the disease under study within 2 weeks prior to apheresis(or within five half-lives of the drug, whichever is shorter), including but not limited to cytotoxic therapy, proteasome inhibitors, immunomodulators, targeted therapy, radiotherapy, epigenetic therapy, etc.; Received anti-PD-1/PD-L1 monoclonal antibody or other investigational drug/invasive medical device within 4 weeksprior to apheresis;
11. Vaccination with live attenuated vaccine or mRNA vaccine within 8 weeks and inactivated vaccine within 4 weeks before screening;
12. Patients who are allergic or intolerant to CLD drugs, tocilizumab, or allergic to the ingredients of CT071 cell infusion preparation (DMSO); Or previous history of other severe allergies, such as anaphylactic shock;
13. Positive test results for any of the following: human immunodeficiency virus (HIV) antibody, Treponema pallidum antibody, hepatitis C virus (HCV) RNA, hepatitis B virus (HBV) surface antigen (HBsAg), HBV DNA;
14. The toxicities caused by the previous treatment have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1, except for alopecia and other tolerable events as judged by the investigator;
15. Left ventricular ejection fraction (LVEF) < 50%;
16. Oxygen saturation < 92% at room air;
17. Received glucocorticoids within 7 days prior to apheresis, with the exception of inhaled glucocorticoids and physiologic replacement doses;
18. Other conditions considered inappropriate for participation in this clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
DLT after CT071 infusion | Assessed from the date of first dose of study treatment until 21~28 days
  Evaluate DLT and adverse events after CT071 infusion
AE of Neurotoxicity and cytokine release syndrome after CT071 infusion | From first dose of study drug adminisration to end of treatment (up to 12 months)
  Cytokine release syndrome（CRS）should be evaluated according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading，higher scores mean a worse outcome.
Adverse Events (AE) after CT071 infusion | From first dose of study drug administration to end of treatment (up to 12 months)
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), with the exception of cytokine release syndrome (CRS), and immune effector cellassociated neurotoxicity syndrome (ICANS).

SECONDARY OUTCOMES:
Level of CAR-T Cell Expansion (proliferation), and Persistence | From first dose of study drug administration to 26 weeks
  Levels of cell expansion (proliferation), and persistence via monitoring CAR-T positive cell counts and CAR transgene level will be reported.
Cytokines in the peripheral blood after CT071 infusion | From first dose of study drug administration to 4 weeks
  Serum concentrations of interleukin (IL)-2, IL-6，IL-8，IL-10，interferon-gamma (IFN-γ), and TNF-α after CT071 infusion
Preliminary evaluation of immunogenicity | From first dose of study drug administration to end of treatment (up to 12 months)
  ADA positive rate
Overall response rate (ORR) as measured by International Myeloma Working Group (IMWG) criteria after CT071 infusion | From first dose of study drug administration to end of treatment (up to 12 months)
  ORR defined as proportion of patients achieving PR or better based on IMWG defined response criteria
Rate of very good partial response (VGPR) and above, complete response/stringent complete response (CR/sCR); | From first dose of study drug administration to end of treatment (up to 12 months)
  Rate of very good partial response (VGPR) and above defined as proportion of patients achieving VGPR or better based on IMWG defined response criteria;
  Rate of complete response/stringent complete response (CR/sCR) defined as proportion of patients achieving CR or better based on IMWG defined response criteria.
Duration of response (DOR) | From first dose of study drug administration to end of treatment (up to 12 months)
  DOR is defined as the time from first achieving PR or better to confirmed disease progression or death from any cause.
Minimal residual disease (MRD) negative rate; | From first dose of study drug administration to end of treatment (up to 12 months)
  Minimal residual disease (MRD) negative rate is defined as the proportion of patients with VGPR or better who achieved 10-5 sensitivity of nucleated cell.
Time to response (TTR) | From first dose of study drug administration to end of treatment (up to 12 months)
  TTR defined as the time from the date of apheresis to the date of initial assessment of PR or better in patients with a best response assessment of partial response or better according to IMWG2016 criteria.
Progression-free survival (PFS) | From first dose of study drug administration to end of treatment (up to 12 months)
  PFS defined as the time from the date of apheresis of the subject to the first assessment of confirmed disease progression or death from any cause according to IMWG2016 criteria, whichever occurs first.
Overall survival (OS) | From first dose of study drug administration to death
  OS defined as the time from the date of apheresis of the subject to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

REFERENCES:
- [Derived] Jin L, Gu S, Ruan Q, Lu J, Qiang W, He H, Fan X, Liu J, Guo P, Meng X, Rajakumaraswamy N, Chen D, Li Z, Du J. GPRC5D-targeted CAR T-cell therapy (CT071) in patients with relapsed or refractory multiple myeloma: a first-in-human, single-centre, single-arm, phase 1 trial. Lancet Haematol. 2025 Oct;12(10):e798-e807. doi: 10.1016/S2352-3026(25)00176-0. PMID 41062204